CLINICAL TRIAL: NCT01253343
Title: Salivary Hormones and Pediatric Aggression and Violence: A Feasibility Study
Brief Title: Pediatric Aggression and Violence
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0892
Record Dates: First submitted 2010-11-01; First posted 2010-12-03 (Estimated); Results first posted 2013-08-28 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-05

CONDITIONS: Pediatric Aggression and Violence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva specimens will be retained for future research use for particpants who have given proper consent.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- inpatient high aggression
- inpatient low aggression

SUMMARY:
Violence and aggression on pediatric psychiatry units has led to staff and patient injuries and even deaths around the country. In an effort to improve safety, the investigators have developed a method (with the Brief Rating of Child and Adolescent Aggression) of identifying children and adolescents at a higher risk for aggression and violence on the units. In order to improve this prediction, the investigators plan to study salivary hormones in low risk children and high risk children. The salivary hormones to be studied include cortisol, testosterone, and dehydroepiandrosterone sulfate (DHEAS). The investigators expect to improve the investigators current ability to predict the severity and type of pediatric aggression and violence on the inpatient units by combining information from the Brief Rating of Child and Adolescent Aggression (BRACHA), the Predatory-Affective Aggression Scale (Vitiello et al., 1990), and salivary hormones.

ELIGIBILITY:
Inclusion Criteria:

1. Prepubescent males (per parent report), African American or Caucasian, between 7 and 9 years old
2. Ability of the subject to provide assent
3. Ability of the guardian to give parental permission
4. Completion of the BRACHA questionnaire
5. Completion of the Predatory-Affective Aggression Scale (PAAS)

Exclusion Criteria:

1. Viral or bacterial infection or treatment with antibiotics within two weeks of screening
2. Recent surgery (within 8 weeks of screening)
3. Bleeding gums (within 8 weeks of screening)
4. Currently detained in a juvenile detention
5. Currently taking medications such as antipsychotic medications (besides Aripiprazole), steroids and beta adrenergic agonists that affect hormones
6. If it is the investigator's clinical judgment that the subject should be excluded if it is in the subject's best interest or due to any other factor that may interfere with study results

Ages: 7 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 24 male subjects (ages 7-11) will be recruited to two groups from inpatient units at CCHMC:
  1. Inpatient high aggression: Twelve inpatient males (6 African-American and 6 Caucasian) will be recruited based on completion of the BRACHA and the Predatory-Affective Aggression Scale.
  2. Inpatient low aggression: Twelve inpatient males (6 African-American and 6 Caucasian) will be recruited based on completion of the BRACHA and the Predatory-Affective Aggression Scales.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Childrens Hospital, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2011 and November 2011, we recruited 17 psychiatrically hospitalized boys (ages 7 to 9 years). We categorized the 17 participants into 2 groups, high aggression risk and low aggression risk, based on their initial BRACHA score.
Pre-assignment Details: Inclusion criteria included boys aged 7 to 9 years, with BRACHA scores, admitted to a psychiatric inpatient unit. Exclusion criteria included presence of infection requiring antibiotics within 2 weeks, recent surgery within 8 weeks, bleeding gums within 8 weeks of admission, current detainment in juvenile detention, and steroid use.
Groups:
- Inpatient High Aggression: The high- risk group was defined as having a BRACHA score >7.5.
- Inpatient Low Aggression: The low- risk group was defined as having a BRACHA score <7.5.
Period: Overall Study
Arm/Group | Inpatient High Aggression | Inpatient Low Aggression
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inpatient High Aggression: The high- risk group was defined as having a BRACHA score ≥ 8.
- Inpatient Low Aggression: The low- risk group was defined as having a BRACHA score ≤6.5.
- Total: Total of all reporting groups
Arm/Group | Inpatient High Aggression | Inpatient Low Aggression | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 8 | 17
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8 (1) | 8 (1) | 8 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Salivary Hormone Correlation With Brief Rating of Aggression by Children and Adolescent (BRACHA) Score
Description: We collected three saliva samples from each participant over a 24-hour period on one of the initial three hospital days to determine the peripheral concentrations of cortisol, dehydroepiandrosterone (DHEA), and testosterone. We then compared these levels with the participants BRACHA score. We wanted to determine if hormone concentrations could improve the BRACHA's accuracy of predicting pediatric aggression during psychiatric hospitalization.
Time Frame: Collected on one or two days
Population: The number of participants for analysis was supposed to be 24 based on Kelsey's sample size calculation (Kelsey et al., Methods in Observational Epidemiology, 2nd Edition, Table 12-15). However, due to funding constraints we only collected samples from 17 participants.
Measure: Mean (Standard Deviation); unit: ul/dL
Groups:
- Low Aggression Group + Cortisol Sample1: Low Aggression= BRACHA Score <7.5 Saliva Sample 1 was obtained immediately upon awaking before eating or teeth brushing
- Low Aggression Group + Cortisol Sample2: Low Aggression= BRACHA Score <7.5 Saliva Sample 2 was obtained 28-30 minutes after Sample 1
- Low Aggression Group + Cortisol Sample3: Low Aggression= BRACHA Score <7.5 Saliva Sample 3 was obtained between 3:45pm and 7:45 pm, depending on when the participant last ate food.
- High Aggression Group + Cortisol Sample1: High Aggression= BRACHA Score >7.5 Saliva Sample 1 was obtained immediately upon awaking before eating or teeth brushing
- High Aggression Group + Cortisol Sample2: High Aggression= BRACHA Score >7.5 Saliva Sample 2 was obtained 28-30 minutes after Sample 1
- High Aggression Group + Cortisol Sample3: High Aggression= BRACHA Score >7.5 Saliva Sample 3 was obtained between 3:45pm and 7:45 pm, depending on when the participant last ate food.
Arm/Group | Low Aggression Group + Cortisol Sample1 | Low Aggression Group + Cortisol Sample2 | Low Aggression Group + Cortisol Sample3 | High Aggression Group + Cortisol Sample1 | High Aggression Group + Cortisol Sample2 | High Aggression Group + Cortisol Sample3
Number analyzed (Participants) | 8 | 6 | 6 | 9 | 9 | 9
ul/dL | 0.8 (0.9) [2 to 3] | 0.4 (0.1) [2 to 3] | 0.3 (0.3) | 0.4 (0.2) | 0.8 (0.3) | 0.2 (0.1)

2. Primary Outcome: Salivary Hormone Correlation With Brief Rating of Aggression by Children and Adolescent (BRACHA) Score.
Description: as for outcome 1
Time Frame: Collected on one or two days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Low Aggression Group + DHEA Sample1; Low Aggression Group + TestosteroneSample1: Low Aggression= BRACHA Score <7.5 Saliva Sample 1 was obtained immediately upon awaking before eating or teeth brushing
- Low Aggression Group + DHEA Sample2; Low Aggression Group + TestosteroneSample2: Low Aggression= BRACHA Score <7.5 Saliva Sample 2 was obtained 28-30 minutes after Sample 1
- Low Aggression Group + DHEA Sample3; Low Aggression Group + TestosteroneSample3: Low Aggression= BRACHA Score <7.5 Saliva Sample 3 was obtained between 3:45pm and 7:45 pm, depending on when the participant last ate food.
- High Aggression Group + DHEASample1; High Aggression Group + TestosteroneSample1: High Aggression= BRACHA Score >7.5 Saliva Sample 1 was obtained immediately upon awaking before eating or teeth brushing
- High Aggression Group + DHEASample2; High Aggression Group + TestosteroneSample2: High Aggression= BRACHA Score >7.5 Saliva Sample 2 was obtained 28-30 minutes after Sample 1
- High Aggression Group + DHEASample3; High Aggression Group + TestosteroneSample3: High Aggression= BRACHA Score >7.5 Saliva Sample 3 was obtained between 3:45pm and 7:45 pm, depending on when the participant last ate food.
Arm/Group | Low Aggression Group + DHEA Sample1 | Low Aggression Group + DHEA Sample2 | Low Aggression Group + DHEA Sample3 | Low Aggression Group + TestosteroneSample1 | Low Aggression Group + TestosteroneSample2 | Low Aggression Group + TestosteroneSample3 | High Aggression Group + DHEASample1 | High Aggression Group + DHEASample2 | High Aggression Group + DHEASample3 | High Aggression Group + TestosteroneSample1 | High Aggression Group + TestosteroneSample2 | High Aggression Group + TestosteroneSample3
Number analyzed (Participants) | 8 | 6 | 6 | 8 | 6 | 6 | 9 | 9 | 9 | 9 | 9 | 9
pg/mL | 85.7 (30.9) | 121.1 (64.4) | 111.9 (45.8) | 37.3 (8.2) | 38.8 (16.5) | 42.7 (14.4) | 97.3 (95.1) | 132.3 (101.6) | 95.5 (58.2) | 45.1 (25.8) | 46.9 (17.8) | 37 (12.5)

ADVERSE EVENTS:
Time Frame: 6 months
Description: No AEs were reported. This was a less than minimal risk study. The saliva collection was the only procedure conducted and is non-invasive.
Arm/Group | Inpatient High Aggression | Inpatient Low Aggression
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes